CLINICAL TRIAL: NCT04418180
Title: Fenofibrate as an Adjuvant to Phototherapy in Pathological Unconjugated Hyperbilirubinemia in Full Term Infants: A Randomized Control Trial.
Brief Title: Fenofibrate Therapy in Pathological Unconjugated Hyperbilirubinemia in Full Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abd Elazeez Attala Shabaan, Professor, Mansoura University
Other Study IDs: MansouraU003
Record Dates: First submitted 2020-05-29; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Neonatal Jaundice
Keywords: Fenofibrate, Neonatal hyperbilirubinemia, Phototherapy
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia, Neonatal | interventions — Fenofibrate

ARMS (3):
- GROUP1 (Active Comparator): group receiving single dose fenofibrate
  Interventions: Drug: Fenofibrate
- GROUP2 (Active Comparator): group receiving double dose fenofibrate
  Interventions: Drug: Fenofibrate
- GROUP3 (Placebo Comparator): photo therapy only
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenofibrate — Patients were randomly assigned to receive oral fenofibrate 10 mg/kg/hr
  Arms: GROUP1; GROUP2
Drug: Placebo — oral distilled water
  Arms: GROUP3

SUMMARY:
Background: Despite widespread phototherapy usage, many newborn infants remain in need of other lines of invasive therapy such as intravenous immunoglobulins and exchange transfusions.

Objective: To assess the efficacy and the safety of adding fenofibrate to phototherapy for treatment of pathological jaundice in full term infants.

Design/Methods: We conducted a double blinded randomized control study on 180 full-term infants with pathological unconjugated hyperbilirubinemia admitted to the NICU of Mansoura University Children's Hospital. They were randomly assigned to receive either oral fenofibrate 10 mg /kg /day for one day or two days or placebo. Primary outcome was total serum bilirubin values after 12, 24, 36, 48 hours from intervention. Secondary outcomes were total duration of treatment, need for exchange transfusions and intravenous immunoglobulin, exclusive breast-feeding on discharge, and adverse effects of fenofibrate.

ELIGIBILITY:
Inclusion Criteria:

* we included appropriate for gestational age full-term infants with pathological unconjugated hyperbilirubinemia who are candidate for phototherapy according to American academy of pediatrics guidelines

Exclusion Criteria:

* Full term infants with intrauterine growth restriction, congenital malformations, conjugated hyperbilirubinemia, severe jaundice initially required exchange transfusion, skin abrasions or infection, and preterm infants were excluded

Max Age: 28 Days | Sex: All
Age Groups: Child
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Total serum bilirubin | 24 hours of treatment
  measure level of serum total bilirubin (mg/dl)
Total serum bilirubin | 48 hours of treatment
  measure level of serum total bilirubin (mg/dl)
Total serum bilirubin | 72 hours of treatment
  measure level of serum total bilirubin (mg/dl)

SECONDARY OUTCOMES:
length of hospital stay | expected 3 days of treatment
  Duration of hospital admission (days)
duration of photo therapy | expected 48 hours of treatment
  duration of photo therapy (hours)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Awad MH, Amer S, Hafez M, Nour I, Shabaan A. "Fenofibrate as an adjuvant to phototherapy in pathological unconjugated hyperbilirubinemia in neonates: a randomized control trial.". J Perinatol. 2021 Apr;41(4):865-872. doi: 10.1038/s41372-020-00861-2. Epub 2020 Oct 17. PMID 33070152